CLINICAL TRIAL: NCT05423041
Title: Prospective Clinical Trial Designed to Evaluate the Repeatability and Reproducibility of the Intelon BOSS(tm) System
Brief Title: A Prospective Clinical Trial Designed to Evaluate the Repeatability and Reproducibility of the Intelon BOSS(tm) System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intelon Optics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P22-01
Record Dates: First submitted 2022-06-08; First posted 2022-06-21 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2022-09

CONDITIONS: Corneal Transplant; Corneal Crosslinking; Healthy Eyes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Biomechanical Imaging of the Eye (Other)
  Interventions: Diagnostic Test: BOSS Imaging

INTERVENTIONS:
Diagnostic Test: BOSS Imaging — Biomechanical Imaging of Cornea and Lens

SUMMARY:
This is a prospective, open-label, single-site clinical trial designed to evaluate the repeatability and reproducibility of biomechanical imaging by the updated version of the BOSS device. Subjects will undergo unilateral biomechanical mapping of the cornea and lens by three (3) BOSS devices operated by three (3) different operators.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older

Exclusion Criteria:

* No light perception
* Any systemic disease or disorder which would prohibit image aquisition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-05-14 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

PRIMARY OUTCOMES:
Analysis of variance in BOSS analysis to determine repeatability and reproducibility | 30 days
  A random effect model will be used to assess variation due to device/operator configuration

CONTACTS AND LOCATIONS:
Locations (1):
- Vold Vision plc, Fayetteville, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No